CLINICAL TRIAL: NCT03637491
Title: A PHASE 1B/2 STUDY TO EVALUATE SAFETY AND CLINICAL ACTIVITY OF COMBINATIONS OF AVELUMAB, BINIMETINIB AND TALAZOPARIB IN PATIENTS WITH LOCALLY ADVANCED OR METASTATIC RAS-MUTANT SOLID TUMORS
Brief Title: A Study of Avelumab, Binimetinib and Talazoparib in Patients With Locally Advanced or Metastatic RAS-mutant Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Available clinical data has shown limited anti-tumor activity and reaching target study drug dose levels may not be feasible.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: B9991033; 2018-000124-34 (EudraCT Number)
Record Dates: First submitted 2018-08-10; First posted 2018-08-20 (Actual); Results first posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-12

CONDITIONS: Pancreatic Cancer
Keywords: KRAS; NRAS; PDAC; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — avelumab; binimetinib; talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Avelumab and binimetinib (Experimental): Open label
  Interventions: Drug: Avelumab; Drug: Binimetinib
- Avelumab, binimetinib and talazoparib (Experimental): Open label
  Interventions: Drug: Avelumab; Drug: Binimetinib; Drug: Talazoparib
- Binimetinib and talazoparib. (Experimental): Open label.
  Interventions: Drug: Binimetinib; Drug: Talazoparib

INTERVENTIONS:
Drug: Avelumab — IV treatment
  Other Names: MSB0010718C
  Arms: Avelumab and binimetinib; Avelumab, binimetinib and talazoparib
Drug: Binimetinib — Oral treatment
  Other Names: MEK162; ARRY-438162
Drug: Talazoparib — Oral treatment
  Other Names: MDV3800, BMN 673
  Arms: Avelumab, binimetinib and talazoparib; Binimetinib and talazoparib.

SUMMARY:
This Phase 1b/2 study will examine the effects of the study drugs, avelumab, binimetinib and talazoparib when given in a 2 (doublet) or 3 (triplet) drug combination, in patients with locally advanced or metastatic RAS-mutant solid tumors. The Phase 1b part of the study will assess if the different study drugs can be given together safely and which doses to use for further research. Phase 2 will test if the study treatments have an effect on tumor size and growth, and gather more information about potential side effects.

DETAILED DESCRIPTION:
This is a Phase 1b/2, open label, multi-center, safety, clinical activity, pharmacokinetic (PK), and pharmacodynamics (PD) study of combinations of avelumab, binimetinib and talazoparib in adult patients with metastatic pancreatic ductal adenocarcinoma and other locally advanced or metastatic KRAS- or NRAS-mutant solid tumors.

The Phase 1b part of this study will initially assess doublet drug combinations to determine a recommended dose for further investigation. Following this, the recommended dose for the combination of avelumab, binimetinib and talazoparib (triplet) will be determined. The recommended doses for the doublet and triplet combinations will be used in the Phase 2 part of the study, which will assess the safety and preliminary anti-tumor activity of the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of locally advanced (primary or recurrent) or metastatic solid tumors that are not amenable for treatment with curative intent as follows:

  1. Metastatic pancreatic ductal adenocarcinoma; or
  2. Phase 2 only: Stage IIIb/IV NSCLC or other advanced solid tumors with documented positive KRAS or NRAS mutation as determined using a validated test performed in a CAP/CLIA-certified laboratory (or other comparable local or regional certification).
* Have had disease progression during or following at least 1 and not more than 2 prior lines of treatment for advanced or metastatic disease.
* Patients with NSCLC must have previously received treatment with an anti-PD-1 or anti-PD-L1 agent for advanced disease.
* Measurable disease as per RECIST v1.1 criteria.
* Provision of a baseline tumor sample.
* Age ≥18 years (Japanese patients must be ≥20 years old)
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
* Adequate bone marrow, renal and liver functions.
* Adequate cardiac function.
* Informed consent provided.

Exclusion Criteria:

* Prior treatment with avelumab, a PARP inhibitor or MEK inhibitor.
* Prior systemic anti-cancer therapy within 2 weeks prior to study enrollment.
* Persisting toxicity related to prior therapy.
* Current use of immunosuppressive medication.
* Known history of immune-mediated colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis, uveitis or iritis.
* Active or prior autoimmune disease that might deteriorate when receiving an immunostimulatory agent.
* Diagnosis of myelodysplastic syndrome (MDS).
* Known symptomatic brain metastases requiring steroids.
* Known history of testing positive for HIV or hepatitis.
* Clinically significant (ie, active) cardiovascular disease.
* History of thromboembolic or cerebrovascular events.
* Current or anticipated use of a P-gp inhibitor, inducer, or inhibitor of breast cancer resistance protein (BCRP)
* Uncontrolled hypertension.
* Concurrent neuromuscular disorder that is associated with the potential of elevated creatinine kinase.
* Known history of Gilbert's syndrome.
* History or current evidence of retinal degenerative disease, retinal vein occlusion (RVO) or current risk factors for RVO.
* Other acute or chronic medical or psychiatric condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (11):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - California Cancer Associates for Research and Excellence, Inc (cCARE), Encinitas, California
  - University of Colorado Denver CTO (CTRC), Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Horizon Oncology Research, LLC, Lafayette, Indiana
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Hospital, Salt Lake City, Utah
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - UZ Gent, Ghent
- Singapore (5):
  - Singapore National Eye Centre, Singapore
  - Singapore General Hospital, Singapore
  - SingHealth Investigational Medicine Unit, Singapore
  - National Heart Centre Singapore, Singapore
  - National Cancer Centre Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Rodon Ahnert J, Tan DS, Garrido-Laguna I, Harb W, Bessudo A, Beck JT, Rottey S, Bahary N, Kotecki N, Zhu Z, Deng S, Kowalski K, Wei C, Pathan N, Laliberte RJ, Messersmith WA. Avelumab or talazoparib in combination with binimetinib in metastatic pancreatic ductal adenocarcinoma: dose-finding results from phase Ib of the JAVELIN PARP MEKi trial. ESMO Open. 2023 Aug;8(4):101584. doi: 10.1016/j.esmoop.2023.101584. Epub 2023 Jun 26. PMID 37379764
- [Derived] Sun C, Fang Y, Labrie M, Li X, Mills GB. Systems approach to rational combination therapy: PARP inhibitors. Biochem Soc Trans. 2020 Jun 30;48(3):1101-1108. doi: 10.1042/BST20191092. PMID 32379297
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991033

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty six participants were screened and 36 were enrolled, one was not treated. This study was planned to included 2 periods: phase 1b and phase 2. Due to the early termination of this study, only the doublet combinations (avelumab + binimetinib and binimetinib + talazoparib) in Phase 1b to find a safe dose were conducted, and neither the triplet combination of Phase 1b nor Phase 2 was initiated.
Groups:
- Avelumab+Binimetinib 30mg (Phase 1b): Avelumab was administered at a fixed dose of 800 mg every 2 weeks (Q2W) in combination with binimetinib at 30 mg twice daily (BID) orally on a continuous daily dosing schedule.
- Avelumab+Binimetinib 45mg (Phase 1b): Avelumab was administered at a fixed dose of 800 mg Q2W in combination with binimetinib at 45 mg BID orally on a continuous daily dosing schedule.
- Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b): Binimetinib 30 mg was administered orally BID (7 days on / 7 days off) with talazoparib at 0.75 mg once daily (QD) orally on a continuous dosing schedule.
- Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b): Binimetinib 45 mg was administered orally BID (7 days on / 7 days off) with talazoparib at 0.75 mg once daily (QD) orally on a continuous dosing schedule.
Period: Overall Study
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b)
Started | 10 | 12 | 7 | 6
Received Treatment | 10 | 12 | 7 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 10 | 12 | 7 | 6
Not completed — Death | 9 | 9 | 5 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Study Terminated By Sponsor | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Avelumab+Binimetinib 30mg (Phase 1b): Avelumab was administered at a fixed dose of 800 mg Q2W in combination with binimetinib at 30 mg BID orally on a continuous daily dosing schedule.
- Total: Total of all reporting groups
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b) | Total
Number analyzed (Participants) | 10 | 12 | 7 | 6 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.30 (11.10) | 65.25 (8.56) | 68.57 (9.61) | 68.00 (9.94) | 66.40 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 6 | 3 | 16
  Male | 6 | 9 | 1 | 3 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 12 | 5 | 5 | 32
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 0 | 1
  White | 9 | 12 | 6 | 5 | 32
  Not Reported | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) During the Primary DLT Evaluation Period (Cycle 1) in Phase 1b
Description: Any adverse events (AEs) occurring in the first cycle of treatment (28 days) which were attributable to study drugs and met DLT criteria. DLT was defined as hematologic: Grade 4 neutropenia lasting>5 days; febrile neutropenia; neutropenic infection; Grade >=3 thrombocytopenia with bleed; Grade 4 thrombocytopenia; Grade 4 anemia; non-hematologic: Grade ≥3 toxicities (with some exceptions) ; Grade≥3 creatinine phosphokinase (CPK) with creatinine >= 1.5xbaseline; Grade 3 troponin increase with cardiac toxicity; potential Hy's Law cases; eye disorders: retinopathy or retinal detachment Grade≥3; retinal vascular disorder; Grade≥3 uveitis, blurred vision, flashing lights, floaters or others for >21 consecutive days; other Grade 4; cardiac disorders: absolute LVEF decrease >10% and the LVEF was below LLN; other Grade≥3; respiratory disorders: interstitial lung disease Grade≥2; bronchospasm Grade 3; skin and subcutaneous tissue disorders; non-adherence to treatment schedule; dose reductions.
Time Frame: From date of first study treatment to day 28 of study treatment (Up to 28 days)
Population: The safety analysis set included all enrolled participants who receive at least 1 dose of study treatment. The DLT-evaluable analysis set was a subset of the safety analysis set and included all enrolled participants in Phase 1b who were eligible for the study, received at least one dose of the combination treatment, and either experienced DLT during the first cycle (28 days) of treatment, or completed the DLT observation period for the first cycle of treatment without DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b)
Number analyzed (Participants) | 10 | 11 | 6 | 5
Participants | 3 | 5 | 2 | 2

2. Primary Outcome: Phase 2: Confirmed Objective Response (OR) Based on Investigator Assessment Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Description: Confirmed OR, defined as a complete response (CR) or partial response (PR) per RECIST v1.1. CR was defined as complete disappearance of all target and non-target lesions, with the exception of nodal disease and sustained for at least 4 weeks. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 mm. PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions. Both CR and PR must be confirmed by repeated assessments performed no less than 4 weeks after the criteria for response were first met.
Time Frame: From date of first study treatment until the date of first documentation of progressive disease or death due to any cause (assessed for a maximum duration of up to 31 months).
Population: Due to the early termination of this study, Phase 2 was not initiated and therefore no Phase 2 efficacy results were collected and summarized.
Groups:
- Avelumab Binimetinib and Talazoparib: Since phase 2 was not initiated, the dose and details of arm haven't been confirmed.
Arm/Group | Avelumab Binimetinib and Talazoparib
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Adverse Events During the On-Treatment Period
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent adverse event (TEAE) means event between first dose of study treatment and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. An SAE was an AE resulting in any of death; inpatient hospitalization; life-threatening experience; disability; congenital anomaly or deemed significant for any other reason. Symptoms of infusion-related reactions (IRRs) may include, but were not limited to, fever, chills, flushing, hypotension, dyspnea, wheezing, back pain, abdominal pain, and urticaria. Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: From the first dose of study treatment through minimum (30 days + last dose of study treatment, start day of new anti-cancer drug therapy - 1 day) assessed for a maximum duration of up to 31 months
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b)
Number analyzed (Participants) | 10 | 12 | 7 | 6
Participants
  participants with TEAEs | 10 | 12 | 7 | 6
  participants with grade ≥ 3 TEAEs | 10 | 9 | 4 | 5
  participants with treatment-related TEAEs | 10 | 12 | 7 | 6
  participants with grade ≥ 3 treatment-related TEAEs | 8 | 4 | 0 | 3
  participants with serious TEAEs | 6 | 9 | 3 | 3
  participants with serious treatment-related TEAEs | 2 | 1 | 0 | 2
  participants with TEAEs leading to discontinuation of Avelumab | 1 | 2 | 0 | 0
  participants with TEAEs leading to discontinuation of Binimetinib | 3 | 4 | 1 | 2
  participants with TEAEs leading to discontinuation of Talazoparib | 0 | 0 | 1 | 2
  participants with TEAEs leading to discontinuation of any study drug | 3 | 4 | 1 | 2
  participants with TEAEs leading to discontinuation of all study drugs | 1 | 1 | 1 | 0
  participants with treatment-related TEAEs leading to discontinuation of Avelumab | 1 | 1 | 0 | 0
  participants with treatment-related TEAEs leading to discontinuation of Binimetinib | 3 | 3 | 0 | 1
  participants with treatment-related TEAEs leading to discontinuation of Talazoparib | 0 | 0 | 0 | 1
  participants with treatment-related TEAEs leading to discontinuation of any study drug | 3 | 3 | 0 | 1
  participants with treatment-related TEAEs leading to discontinuation of all study drugs | 1 | 0 | 0 | 0
  participants with TEAEs leading to death | 0 | 3 | 2 | 1
  participants with treatment-related TEAEs leading to death | 0 | 0 | 0 | 0
  participants with infusion-related reactions (IRRs) | 3 | 1 | 0 | 0

4. Secondary Outcome: Number of Participants With Hematology Laboratory Abnormalities During the On-Treatment Period Graded by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE), Version 4.03
Description: Laboratory abnormalities were graded by NCI CTCAE version 4.03. Anemia, hemoglobin increased, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, white blood cell decreased were evaluated. This outcome measure calculated the number of participants with laboratory abnormalities whose maximum on-treatment CTCAE Grade were 1-4.
Time Frame: Prior to study drug administration on Days 1 and 15 of each treatment cycle, until 30 days after last dose (assessed for a maximum duration of up to 31 months)
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b)
Number analyzed (Participants) | 10 | 12 | 7 | 6
Participants
  ANEMIA | 9 | 9 | 7 | 5
  HEMOGLOBIN INCREASED | 0 | 0 | 1 | 0
  LYMPHOCYTE COUNT DECREASED | 6 | 7 | 5 | 6
  LYMPHOCYTE COUNT INCREASED | 1 | 1 | 0 | 0
  NEUTROPHIL COUNT DECREASED | 0 | 1 | 1 | 2
  PLATELET COUNT DECREASED | 3 | 3 | 4 | 3
  WHITE BLOOD CELL DECREASED | 2 | 2 | 0 | 4

5. Secondary Outcome: Number of Participants With Chemistry Laboratory Abnormalities During the On-Treatment Period Graded by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE), Version 4.03
Description: Laboratory abnormalities were graded by NCI CTCAE version 4.03. Alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, creatine phosphokinase (cpk) increased, creatinine increased, gamma-glutamyl transferase (ggt) increased, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, hypophosphatemia, lipase increased, serum amylase increased were evaluated. This outcome measure calculated the number of participants with laboratory abnormalities whose maximum on-treatment CTCAE Grade were 1-4.
Time Frame: as for outcome 4
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b)
Number analyzed (Participants) | 10 | 12 | 7 | 6
Participants
  ALANINE AMINOTRANSFERASE INCREASED | 5 | 5 | 3 | 2
  ALKALINE PHOSPHATASE INCREASED | 9 | 7 | 6 | 5
  ASPARTATE AMINOTRANSFERASE INCREASED | 8 | 8 | 6 | 3
  BLOOD BILIRUBIN INCREASED | 4 | 0 | 0 | 1
  CPK INCREASED | 6 | 7 | 3 | 1
  CREATININE INCREASED | 8 | 11 | 6 | 4
  GGT INCREASED | 8 | 4 | 6 | 2
  HYPERCALCEMIA | 2 | 1 | 1 | 0
  HYPERGLYCEMIA | 5 | 6 | 4 | 5
  HYPERKALEMIA | 1 | 3 | 1 | 0
  HYPERMAGNESEMIA | 0 | 0 | 0 | 0
  HYPERNATREMIA | 0 | 0 | 0 | 1
  HYPOALBUMINEMIA | 7 | 11 | 5 | 3
  HYPOCALCEMIA | 0 | 1 | 0 | 0
  HYPOGLYCEMIA | 2 | 2 | 0 | 1
  HYPOKALEMIA | 4 | 1 | 3 | 3
  HYPOMAGNESEMIA | 3 | 2 | 2 | 1
  HYPONATREMIA | 5 | 4 | 2 | 0
  HYPOPHOSPHATEMIA | 3 | 1 | 1 | 0
  LIPASE INCREASED | 1 | 3 | 0 | 1
  SERUM AMYLASE INCREASED | 2 | 5 | 0 | 0

6. Secondary Outcome: Predose Concentration During Multiple Dosing (Ctrough) for Avelumab
Description: Ctrough was the pre-dose concentration during multiple dosing and was directly observed from data. The lower limit of quantification (LLQ) was 0.20 microgram per milliliter. Concentration values below the LLQ were set to zero. Geometric Mean analysis was on the log scale. Zero values were not included in geometric mean and geometric coefficient of variation calculation. The geometric coefficient of variation is expressed in percentage.
Time Frame: Pre-dose on Day 1, and Day 15 of Cycle 1 (each cycle is 28 days); Day 1 and Day 15 of Cycle 2; and Day 1 of Cycles 3, 5, 9 and 12.
Population: Number of participants analyzed: participants who had at least 1 concentration measurement for avelumab. Therefore, only 2 treatment groups including avelumab were analyzed. Number analyzed: participants who had avelumab concentrations above the LLQ at specific time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (ug/mL)
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b)
Number analyzed (Participants) | 10 | 12
microgram per milliliter (ug/mL)
  CYCLE1_DAY15: number analyzed (Participants) | 9 | 12
  CYCLE1_DAY15 | 22.38 (59) | 28.82 (57)
  CYCLE2_DAY1: number analyzed (Participants) | 7 | 9
  CYCLE2_DAY1 | 29.26 (39) | 38.28 (52)
  CYCLE2_DAY15: number analyzed (Participants) | 5 | 9
  CYCLE2_DAY15 | 40.86 (42) | 37.26 (59)
  CYCLE3_DAY1: number analyzed (Participants) | 1 | 7
  CYCLE3_DAY1 | 31.30 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated. | 34.69 (75)
  CYCLE5_DAY1: number analyzed (Participants) | 1 | 5
  CYCLE5_DAY1 | 28.00 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated. | 36.51 (38)
  CYCLE9_DAY1: number analyzed (Participants) | 0 | 2
  CYCLE9_DAY1 |  | 46.49 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated.
  CYCLE12_DAY1: number analyzed (Participants) | 0 | 2
  CYCLE12_DAY1 |  | 38.77 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated.

7. Secondary Outcome: Predose Concentration During Multiple Dosing (Ctrough) for Binimetinib
Description: Ctrough was directly observed from data. Ctrough = concentration prior to study drug administration. The LLQ was 1.00 ng/mL. Concentration values below the LLQ were set to zero. Geometric Mean analysis was on the log scale. Zero values were not included in geometric mean and geometric coefficient of variation calculation. The geometric coefficient of variation is expressed in percentage.
Time Frame: Predose on Day 15 of Cycle 1 (each cycle is 28 days), Day 1 and Day 15 of Cycle 2, Day 1 of Cycle 3 for avelumab+binimetinib groups, and on Day 8 and Day 15 of Cycle 1, Day 1 of Cycle 2, Day 1 of Cycle 3 for binimetinib+talazoparib groups
Population: Number of participants analyzed: participants who had at least 1 concentration measurement for binimetinib. Number analyzed: participants who had binimetinib concentration values above the LLQ at specific time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b)
Number analyzed (Participants) | 10 | 12 | 7 | 6
ng/mL
  CYCLE1_DAY8: number analyzed (Participants) | 0 | 0 | 2 | 4
  CYCLE1_DAY8 |  |  | 82.90 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated. | 128.6 (49)
  CYCLE1_DAY15: number analyzed (Participants) | 5 | 3 | 1 | 0
  CYCLE1_DAY15 | 87.85 (48) | 88.67 (16) | 22.80 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated. |
  CYCLE2_DAY1: number analyzed (Participants) | 4 | 2 | 0 | 0
  CYCLE2_DAY1 | 55.71 (56) | 107.5 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated. |  |
  CYCLE2_DAY15: number analyzed (Participants) | 3 | 2 | 0 | 0
  CYCLE2_DAY15 | 93.45 (90) | 88.33 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated. |  |
  CYCLE3_DAY1: number analyzed (Participants) | 1 | 1 | 0 | 0
  CYCLE3_DAY1 | 56.60 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated. | 74.90 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated. |  |

8. Secondary Outcome: Predose Concentration During Multiple Dosing (Ctrough) for Talazoparib
Description: Ctrough was directly observed from data. Ctrough = concentration prior to study drug administration. The LLQ was 25 pg/mL. Concentration values below the LLQ were set to zero. Geometric Mean analysis was on the log scale. Zero values were not included in geometric mean and geometric coefficient of variation calculation. The geometric coefficient of variation is expressed in percentage.
Time Frame: Pre-dose on Days 1, 8 and Day 15 of Cycle 1 (each cycle is 28 days), and on Day 1 of Cycle 2 and Cycle 3
Population: Number of participants analyzed: participants who had at least 1 concentration measurement for talazoparib. Therefore, only 2 treatment groups including talazoparib were analyzed. Number analyzed: participants who had talazoparib concentrations above the LLQ at specific time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per millilitre (pg/mL)
Arm/Group | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b)
Number analyzed (Participants) | 7 | 6
picograms per millilitre (pg/mL)
  CYCLE1_DAY8: number analyzed (Participants) | 2 | 4
  CYCLE1_DAY8 | 4856 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated. | 2926 (49)
  CYCLE1_DAY15: number analyzed (Participants) | 1 | 4
  CYCLE1_DAY15 | 5960 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated. | 2683 (65)
  CYCLE2_DAY1: number analyzed (Participants) | 1 | 2
  CYCLE2_DAY1 | 8620 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated. | 2753 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated.
  CYCLE3_DAY1: number analyzed (Participants) | 0 | 1
  CYCLE3_DAY1 |  | 1520 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated.

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Avelumab
Description: Cmax was the maximum observed plasma concentration and was directly observed from data. The LLQ was 0.20 microgram per milliliter. Concentration values below the LLQ were set to zero. Geometric Mean analysis was on the log scale. Zero values were not included in geometric mean and geometric coefficient of variation calculation. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on Day 1, and Day 15 of Cycle 1 (each cycle is 28 days); Day 1 and Day 15 of Cycle 2; and Day 1 of Cycles 3, 5, 9 and 12
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (ug/mL)
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b)
Number analyzed (Participants) | 10 | 12
microgram per milliliter (ug/mL)
  CYCLE1_DAY1: number analyzed (Participants) | 8 | 10
  CYCLE1_DAY1 | 205.3 (22) | 248.6 (14)
  CYCLE1_DAY15: number analyzed (Participants) | 8 | 10
  CYCLE1_DAY15 | 214.2 (20) | 237.4 (45)
  CYCLE2_DAY1: number analyzed (Participants) | 5 | 8
  CYCLE2_DAY1 | 213.0 (20) | 241.5 (26)
  CYCLE2_DAY15: number analyzed (Participants) | 6 | 9
  CYCLE2_DAY15 | 211.5 (17) | 243.0 (19)
  CYCLE3_DAY1: number analyzed (Participants) | 1 | 7
  CYCLE3_DAY1 | 176.0 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated. | 233.7 (28)
  CYCLE5_DAY1: number analyzed (Participants) | 1 | 5
  CYCLE5_DAY1 | 188.0 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated. | 241.9 (21)
  CYCLE9_DAY1: number analyzed (Participants) | 0 | 1
  CYCLE9_DAY1 |  | 257.0 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated.
  CYCLE12_DAY1: number analyzed (Participants) | 0 | 2
  CYCLE12_DAY1 |  | 255.8 (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated.

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Binimetinib
Description: Cmax was the maximum observed plasma concentration and was directly observed from data. The LLQ was 1.00 ng/mL. Concentration values below the LLQ were set to zero. Geometric Mean analysis was on the log scale. Zero values were not included in geometric mean and geometric coefficient of variation calculation. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on Day 1 and Day 8 of Cycle 1
Population: Number of participants analyzed: participants who had at least 1 concentration measurement for binimetinib. Number analyzed: participants who had binimetinib concentrations above the LLQ at specific time point. When Cmax for binimetinib was planned to be evaluated, data collecting for Avelumab+Binimetinib cohort had already been done. Therefore, data of Cmax for binimetinib in Avelumab+Binimetinib groups hadn't been collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b)
Number analyzed (Participants) | 0 | 0 | 7 | 6
ng/mL
  CYCLE1_DAY1: number analyzed (Participants) | 0 | 0 | 5 | 6
  CYCLE1_DAY1 |  |  | 370.24 (64) | 331.74 (63)
  CYCLE1_DAY8: number analyzed (Participants) | 0 | 0 | 4 | 5
  CYCLE1_DAY8 |  |  | 183.53 (180) | 446.81 (59)

11. Secondary Outcome: Number of Participants With Anti-drug Antibody (ADA) Categories
Description: Samples positive for ADA were analyzed for titer. Blood samples were collected for avelumab immunogenicity testing. Treatment-boosted ADA was defined as a positive ADA result at baseline and the titer ≥ 8×baseline titer at least once after treatment with avelumab. Treatment-induced ADA was defined as participants with ADA-negative at baseline and had at least one positive post-baseline ADA result; or if participant did not have a baseline sample, the participant had at least one positive post-baseline ADA result.
Time Frame: from the first dose of study up to Day 1 of Cycle 12 for a maximum of 12 months
Population: Participants in the safety analysis set had at least one ADA/nAb sample collected for avelumab, so only two groups (Avelumab+Binimetinib 30mg [Phase 1b] and Avelumab+Binimetinib 45mg [Phase 1b]) were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b)
Number analyzed (Participants) | 10 | 12
Participants
  ADA never-positive | 8 | 11
  ADA ever-positive | 2 | 1

12. Secondary Outcome: Neutralizing Antibodies (nAb) Against Avelumab
Description: The category of nAb included nAb never-positive, nAb ever-positive, baseline nAb positive, treatment-induced nAb, transient nAb response, persistent nAb response.
Time Frame: from the first dose of study up to Day 1 of Cycle 12 for a maximum of 12 months
Population: Participants in the safety analysis set had at least one ADA/nAb sample collected for avelumab. Due to the low observed immunogenicity rate, nAb analysis was not conducted.
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Percentage of Participants With Confirmed Objective Response (OR) in Phase 1b Based on Investigator Assessment (RECIST v1.1)
Description: OR is defined as complete response (CR) or partial response (PR) according to RECIST v1.1 from the 'start date' (date of first study treatment) until the date of the first documentation of progressive disease (PD). CR was defined as complete disappearance of all target and non-target lesions, with the exception of nodal disease and sustained for at least 4 weeks. PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions. PD was defined as unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy. Both CR and PR must be confirmed by repeat assessments performed no less than 4 weeks after the criteria for response are first met. Clopper-Pearson method was used.
Time Frame: as for outcome 2
Population: The full analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b)
Number analyzed (Participants) | 10 | 12 | 7 | 6
Percentage of participants | 0 [0.0 to 30.8] | 8.3 [0.2 to 38.5] | 0 [0.0 to 41.0] | 0 [0.0 to 45.9]

14. Secondary Outcome: Progression-Free Survival (PFS) Based on Investigator Assessment (RECIST v1.1) in Phase 1b
Description: PFS is defined as the time from the 'start date' (date of first study treatment) to the date of the first documentation of PD or death due to any cause, whichever occurs first. PD was defined as unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy. CIs were calculated using Brookmeyer and Crowley method.
Time Frame: as for outcome 2
Population: The full analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b)
Number analyzed (Participants) | 10 | 12 | 7 | 6
months | 1.7 [1.6 to 2.9] | 3.3 [1.6 to 7.1] | 1.6 [1.0 to 2.3] | 1.8 [1.1 to 4.6]

15. Secondary Outcome: Overall Survival (OS) in Phase 1b
Description: OS is defined as the time from the 'start date' (date of first study treatment) to the date of death due to any cause. CIs were calculated using Brookmeyer and Crowley method.
Time Frame: From date of first study treatment until the date of death due to any cause (assessed for a maximum duration of up to 31 months).
Population: The full analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b)
Number analyzed (Participants) | 10 | 12 | 7 | 6
months | 5.9 [2.9 to 8.6] | 8.0 [3.0 to 20.1] | 2.9 [1.0 to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values, so these summary statistics were not calculated. | 10.7 [1.1 to 10.7]

16. Secondary Outcome: Time-to-Tumor Response (TTR) in Phase 1b
Description: TTR is defined, for patients with an OR, as the time from the 'start date' (date of first study treatment) to the first documentation of objective response (CR or PR) which was subsequently confirmed. OR is defined as complete response (CR) or partial response (PR) according to RECIST v1.1 from the 'start date' until the date of the first documentation of progressive disease (PD). CR was defined as complete disappearance of all target and non-target lesions, with the exception of nodal disease and sustained for at least 4 weeks. PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions. PD was defined as unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy.
Time Frame: as for outcome 2
Population: The full analysis set included all enrolled participants who received at least 1 dose of study treatment and achieved objective response: only 1 participant in the Avelumab+Binimetinib 45mg (Phase 1b) group achieved OR. The summary of this endpoint cannot be estimated due to small sample size (1 participant).
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b)
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Duration of Response (DR) in Phase 1b
Description: DR is defined, for patients with OR, as the time from the first documentation of objective response (CR or PR) to the date of first documentation of PD or death due to any cause. OR is defined as complete response (CR) or partial response (PR) according to RECIST v1.1 from the 'start date' until the date of the first documentation of progressive disease (PD). CR was defined as complete disappearance of all target and non-target lesions, with the exception of nodal disease and sustained for at least 4 weeks. PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions. PD was defined as unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy.
Time Frame: as for outcome 2
Population: as for outcome 16
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b)
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Phase 2: Number of Participants With Programmed Death-Ligand 1 (PD-L1) Expression, DNA Damage Repair (DDR) Gene Alterations, and Tumor Mutational Burden (TMB) in Baseline Tumor Tissue.
Description: PD-L1 expression was defined as the number of PD-L1 positive cells and/or qualitative assessment of PD-L1 staining on tumor and inflammatory cells in regions of interest. DDR gene alterations was defined as the number of somatic and germline mutations present in a panel of genes associated with DDR in baseline tumor derived nucleic acid, in germline nucleic acid and in circulating tumor DNA. TMB was defined as determination/estimation of the frequency of mutations (total and non-synonymous) present in baseline tumor derived nucleic acid samples and in baseline circulating tumor DNA.
Time Frame: Baseline
Population: The biomarkers were for the phase 2 part. since phase 2 was not initiated, the results was not provided.
Arm/Group | Avelumab Binimetinib and Talazoparib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment through minimum (30 days + last dose of study treatment, start day of new anti-cancer drug therapy - 1 day) assessed for a maximum duration of up to 31 months
Arm/Group | Avelumab+Binimetinib 30mg (Phase 1b) | Avelumab+Binimetinib 45mg (Phase 1b) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b)
All-Cause Mortality (participants affected / at risk) | 9/10 | 9/12 | 5/7 | 3/6
Serious Adverse Events (participants affected / at risk) | 6/10 | 9/12 | 3/7 | 3/6
Other Adverse Events (participants affected / at risk) | 10/10 | 12/12 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab+Binimetinib 30mg (Phase 1b) (N=10) | Avelumab+Binimetinib 45mg (Phase 1b) (N=12) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) (N=7) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Chills (General disorders) | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 3 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab+Binimetinib 30mg (Phase 1b) (N=10) | Avelumab+Binimetinib 45mg (Phase 1b) (N=12) | Binimetinib 30mg+Talazoparib 0.75mg (Phase 1b) (N=7) | Binimetinib 45mg+Talazoparib 0.75mg (Phase 1b) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 2 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0
Macular oedema (Eye disorders) | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 2 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 1
Retinopathy (Eye disorders) | 0 | 3 | 0 | 0
Subretinal fluid (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 3 | 4
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 4 | 4 | 2
Fatigue (General disorders) | 2 | 4 | 4 | 1
Mucosal inflammation (General disorders) | 1 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 4 | 1 | 1
Pain (General disorders) | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 2 | 0 | 1
Ammonia increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 3 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 4 | 3 | 0
Blood creatinine increased (Investigations) | 0 | 3 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 2 | 2
Troponin T increased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 3 | 2 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 7 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Diastolic hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 4 | 0 | 1

LIMITATIONS AND CAVEATS:
Because there was a low probability of technical success for achieving target dose levels of the triplet combination while maintaining acceptable tolerability, and only limited anti-tumor activity was observed in this study of participants with mPDAC, a decision on the early termination was made on 14 December 2020. Phase 2 was not initiated, so PD-L1 Expression, DDR Gene Alterations, TMB and OR were not analyzed. Due to the low observed immunogenicity rate, nAb analysis was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT03637491/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT03637491/SAP_001.pdf